CLINICAL TRIAL: NCT05297136
Title: Preoperative Endoscopic Pancreatic Stent to Prevent Pancreatic Fistula After Distal Pancreatectomy: a Randomized Controlled Trial
Brief Title: Preoperative Endoscopic Pancreatic Stent for Distal Pancreatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Yue Sun, Clinical Associate Professor (honorary), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021.728-T
Record Dates: First submitted 2022-03-03; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Pancreatectomy; Pancreatic Fistula
Keywords: Distal Pancreatectomy; Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-op Stenting (Experimental): Pre-operative pancreatic stent inserted by Endoscopic Retrograde Cholangiography, followed by distal pancreatectomy
  Interventions: Procedure: Pancreatic Stenting
- Surgery alone (Active Comparator): Distal pancreatectomy alone
  Interventions: Procedure: No Stent

INTERVENTIONS:
Procedure: Pancreatic Stenting — Pancreatic stent of appropriate size and length is inserted to the pancreatic duct before distal pancreatectomy
  Arms: Pre-op Stenting
Procedure: No Stent — No preoperative stenting with distal pancreatectomy alone
  Arms: Surgery alone

SUMMARY:
Distal pancreatectomy (DP) with or without splenectomy is commonly indicated for pancreatic body or tail lesions. Postoperative pancreatic fistula (POPF) remains the commonest complication after DP. A pre-operatively placed pancreatic stent across papilla can decrease the pressure gradient between pancreatic duct and duodenum. Therefore, the pancreatic juice flow is redirected from the pancreatic transection plane and leakage from pancreatic stump is much reduced. This study aims to evaluate whether pre-operatively placed pancreatic stent can prevent POPF by a randomized controlled trial.

DETAILED DESCRIPTION:
A randomised-controlled trial is performed to evaluate the efficacy of preoperative pancreatic duct stenting in preventing post-operative pancreatic fistula after distal pancreatectomy with or without splenectomy. Patients will be randomised to pre-operative stent group or surgery alone group. Pre-operative pancreatic duct stenting will be performed 1-2 weeks before surgery. The stent will be removed 4 weeks after operation. The post-operative pancreatic fistula rate, morbidity, mortality and total length of stay were compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Elective distal pancreatectomy for primary pancreatic pathology

Exclusion Criteria:

* Informed consent not available
* Emergency distal pancreatectomy
* Presence of pancreatic duct stricture
* Presence of altered anatomy that precludes safe Endoscopic Retrograde Cholangiography (e.g. previous Billroth II gastrectomy)
* History of severe pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative pancreatic fistula | Day 3 after operation
  The number of participants developing post-operative pancreatic fistula, which is defined as drain fluid amylase more than 3 times the upper limit of the normal value of serum amylase on or after postoperative day 3

SECONDARY OUTCOMES:
Number of participants developing post-operative morbidity | 90 days
  Post-operative complications, graded according to the Clavien-Dindo classification, are recorded
Number of participants developing post-operative mortality | 90 days
  All cause mortality after operation was recorded
Total length of hospital stay of participants | 90 days after endoscopy and operation
  The total number of days spent in hospital calculated from the day of admission to discharge for every participant, including the time spent for pre-operative endoscopy and operation
Number of participants developing complications related to Endoscopic Retrograde Cholangiography | 14 days after endoscopy
  All complications occurred after Endoscopic Retrograde Cholangiopancreatography were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Kit Fai Lee, MBBS, Principal Investigator — Clinical Associate Professor (honorary)
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No